CLINICAL TRIAL: NCT02046200
Title: Repositioning Ivermectin for the Treatment of Alcohol Use Disorders
Brief Title: Development of Ivermectin for Alcohol Use Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lara Ray, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IVM; UL1TR000124 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-01-27 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Alcohol Use Disorder
Keywords: ivermectin, alcoholism, alcohol use disorder, treatment
MeSH Terms: conditions — Alcoholism | interventions — Ivermectin; Sugars; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivermectin (Experimental): Ivermectin 30 mg single dose
  Interventions: Drug: Ivermectin; Drug: Alcohol
- Sugar pill (Placebo Comparator): Matched placebo, single dose
  Interventions: Drug: Placebo; Drug: Alcohol

INTERVENTIONS:
Drug: Ivermectin — Ivermectin is a semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum antiparasitic avermectin.
  Other Names: Stromectol
  Arms: Ivermectin
Drug: Placebo — Matched placebo
  Other Names: Sugar pill
  Arms: Sugar pill
Drug: Alcohol
  Other Names: 5% ethanol IV solution

SUMMARY:
Current pharmacotherapies for alcohol use disorders (AUDs) have limited efficacy. Thus, the development of effective treatments for AUDs represents an important public health objective. Repositioning, i.e. using existing approved drugs for other indications, represents a fast and economically feasible approach for drug development. Ivermectin (IVM) is an FDA-approved antiparasitic medication that can significantly reduce alcohol intake in mice, suggesting that it may be useful in the treatment of AUDs in humans. The goal of this project is to provide key clinical evidence that IVM can be repositioned as a novel therapeutic agent to treat AUDs.

DETAILED DESCRIPTION:
Current pharmacotherapies for alcohol use disorders (AUDs) have limited efficacy. Thus, the development of effective treatments for AUDs represents an important public health objective. Repositioning, i.e. using existing approved drugs for other indications, represents a fast and economically feasible approach for drug development. Ivermectin (IVM) is an FDA-approved antiparasitic medication that can significantly reduce alcohol intake in mice, suggesting that it may be useful in the treatment of AUDs in humans. The goal of this project is to provide key clinical evidence that IVM can be repositioned as a novel therapeutic agent to treat AUDs. We will enroll 10 alcohol dependent individuals in a placebo-controlled randomized pilot safety trial of IVM (30 mg orally once) over a 2-day (1-night) inpatient stay at the UCLA CTRC and employ a well-characterized battery of behavioral paradigms (i.e., alcohol administration and cue exposure). The goals of the study are to test: (a) the safety of combining IVM, at a dose currently shown to be safe in humans (30 mg), with moderate doses of alcohol (0.08 g/dl); and (b) whether IVM reduces the reinforcing effects of alcohol during alcohol administration and whether it reduces alcohol craving during cue exposure, as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* age between 21 and 65;
* meet current DSM-V diagnostic criteria for an alcohol use disorder

Exclusion Criteria:

* current treatment for alcohol problems, a history of treatment in the 30 days before enrollment or current treatment seeking;
* a current (last 12 months) DSM-V diagnosis of dependence on any psychoactive substances other than alcohol and nicotine;
* a lifetime DSM-IV diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder;
* positive urine screen for narcotics, amphetamines, or sedative hypnotics;
* serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-R);
* pregnancy, nursing, or refusal to use reliable method of birth control (if female);
* a medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes);
* AST, ALT, or GGT ≥ 3 times upper normal limit;
* currently on prescription medication that contraindicates use of IVN;
* any other circumstances that, in the opinion of the investigators, compromises participant safety.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles; Daniel Roche, PhD, Study Director — University of California, Los Angeles
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UCLA Addictions Laboratory — http://addictions.psych.ucla.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- IVM 30mg First, Then Placebo: First Intervention, Ivermectin (IVM): Single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin.
  Second Intervention, Placebo: Single dose sugar pill, matched to active medication.
- Placebo First, Then IVM 30 mg: First Intervention, Placebo: Single dose sugar pill, matched to active medication.
  Second Intervention, Ivermectin (IVM): Single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin.
Period: First Intervention (1 Day)
Arm/Group | IVM 30mg First, Then Placebo | Placebo First, Then IVM 30 mg
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | IVM 30mg First, Then Placebo | Placebo First, Then IVM 30 mg
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IVM 30mg; Placebo: Ivermectin (IVM): Single dose (30 mg) of a semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin.
  Placebo: Single dose sugar pill matched to active medication.
Arm/Group | IVM 30mg; Placebo
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.82 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Meets criteria for DSM-V AD [Number; unit: participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Heart rate (measured in beats per minute; BPM) will be monitored to determine the safety of combining IVM (30 mg) with moderate doses of alcohol (0.08 g/dl).
  During the infusion, the times for collecting HR will vary based on how long it takes participants to reach the targeted BrACs.
Time Frame: Post-medication administration (hours): 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48; During alcohol infusion at BrAC = 0.00, 0.02, 0.04, 0.06, 0.08 g/dl
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: BPM
Groups:
- Placebo: Single dose sugar pill, matched to active medication.
- IVM 30mg: Ivermectin (IVM): Single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin.
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
BPM
  0 hours post-med | 64.57 (9.74) | 68.36 (20.47)
  0.5 hours post-med | 66.82 (10.91) | 62.82 (11.46)
  1 hour post-med | 66.09 (12.01) | 64.27 (11.60)
  2 hours post-med | 65.18 (13.88) | 61.18 (11.03)
  4 hours post-med | 66.73 (10.60) | 61.55 (12.36)
  6 hours post-med | 63.27 (12.66) | 59.73 (12.62)
  8 hours post-med | 66.36 (13.44) | 62.18 (11.76)
  10 hours post-med | 64.70 (14.33) | 62.64 (10.19)
  12 hours post-med | 72.45 (13.41) | 73.64 (9.31)
  16 hours post-med | 61.18 (12.08) | 58.09 (10.97)
  24 hours post-med | 62.55 (11.09) | 64.64 (10.58)
  48 hours post-med | 69.18 (10.15) | 69.45 (12.49)
  BrAC = 0 | 63.09 (12.69) | 61.00 (11.80)
  BrAC = 0.02 | 67.27 (14.00) | 63.36 (9.00)
  BrAC = 0.04 | 66.91 (10.89) | 61.82 (9.16)
  BrAC = 0.06 | 66.64 (12.83) | 63.09 (9.82)
  BrAC = 0.08 | 66.36 (12.37) | 61.27 (8.21)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.0563, ANOVA

2. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure (measured in mmHg) will be monitored to determine the safety of combining IVM (30 mg) with moderate doses of alcohol (0.08 g/dl).
  Blood pressure is measured at 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post-medication administration; and during alcohol infusion at BrAC = 0.00, 0.02, 0.04, 0.06, 0.08 g/dl. During the infusion, the times for collecting BP will vary based on how long it takes participants to reach the targeted BrACs.
Time Frame: as for outcome 1
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- IVM 30mg: Ivermectin single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin.
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
mmHg
  0 hours post-med | 121 (11.10) | 111.64 (17.35)
  0.5 hours post-med | 118.64 (10.67) | 117 (12.61)
  1 hour post-med | 120.64 (11.44) | 116.27 (11.80)
  2 hours post-med | 121.27 (10.59) | 118.27 (12.48)
  4 hours post-med | 117 (12.15) | 111.91 (12.85)
  6 hours post-med | 117.27 (16.17) | 119.55 (15.33)
  8 hours post-med | 115.18 (13.50) | 107.27 (10.56)
  10 hours post-med | 116.70 (13.49) | 114.09 (13.63)
  12 hours post-med | 116.09 (9.17) | 119.63 (7.99)
  16 hours post-med | 115.64 (17.19) | 115.45 (8.85)
  24 hours post-med | 122 (11.61) | 122.73 (8.72)
  48 hours post-med | 122.72 (8.67) | 121.09 (9.47)
  BrAC = 0 | 120.27 (15.07) | 114.36 (12.75)
  BrAC = 0.02 | 118.55 (10.56) | 114.18 (12.34)
  BrAC = 0.04 | 116.55 (12.36) | 111.27 (10.72)
  BrAC = 0.06 | 112.73 (11.40) | 115.18 (14.08)
  BrAC = 0.08 | 112.45 (12.60) | 108.82 (11.50)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.0342, ANOVA

3. Primary Outcome: Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: as for outcome 1
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
mmHg
  0 hours post-med | 79.64 (10.23) | 75.55 (13.20)
  0.5 hours post-med | 77.45 (11.44) | 75.18 (11.12)
  1 hour post-med | 78.82 (10.30) | 74.91 (10.43)
  2 hours post-med | 79.91 (8.80) | 76.64 (12.14)
  4 hours post-med | 74.55 (10.82) | 72.18 (10.91)
  6 hours post-med | 75.36 (14.49) | 74.55 (11.22)
  8 hours post-med | 72.55 (10.05) | 69.45 (10.46)
  10 hours post-med | 75.30 (11.88) | 73.82 (12.60)
  12 hours post-med | 73.64 (9.84) | 77.27 (6.44)
  16 hours post-med | 72.82 (12.69) | 73.18 (8.81)
  24 hours post-med | 76.09 (12.39) | 78.09 (10.23)
  48 hours post-med | 80.55 (10.96) | 81.55 (10.49)
  BrAC = 0 | 78.18 (11.57) | 74.36 (12.49)
  BrAC = 0.02 | 77.91 (10.01) | 73.73 (10.96)
  BrAC = 0.04 | 77.55 (10.71) | 72.91 (11.89)
  BrAC = 0.06 | 75.27 (9.31) | 74.00 (12.13)
  BrAC = 0.08 | 71.91 (10.90) | 72.73 (10.75)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.1597, ANOVA

4. Primary Outcome: Subjective Effects of Alcohol Using the Alcohol Urge Questionnaire (AUQ)
Description: Subjective effects of alcohol will be measured using the Alcohol Urge Questionnaire (AUQ), which consists of 8 items associated with urge to drink alcohol, rated on a 7 point scale (1 = strongly disagree, 7 = strongly agree).
Time Frame: During alcohol infusion at BrAC = 0.00, 0.02, 0.04, 0.06, 0.08 g/dl period; which is expected to last approximately 6 hours.
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 2.58 (1.74) | 2.90 (2.04)
  BrAC = 0.02 | 3.14 (1.64) | 3.27 (1.65)
  BrAC = 0.04 | 3.02 (1.64) | 3.19 (1.60)
  BrAC = 0.06 | 2.73 (2.00) | 2.60 (1.60)
  BrAC = 0.08 | 2.83 (1.79) | 2.91 (1.87)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.7617, ANOVA

5. Primary Outcome: Subjective Effects of Alcohol Using the Drug Effects Questionnaire (DEQ) - "Feel" Subscale
Description: Subjective effects of alcohol will be measured using the Drug Effects Questionnaire, which consists of 4 items that capture subjective effects, (feeling effects, liking effects, wanting more and being high). The question "Do you feel any drug effects?" was rated on an 11 point scale from 0 to 10 (higher values represent more effects).
Time Frame: as for outcome 4
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 1.36 (2.66) | 0.91 (1.30)
  BrAC = 0.02 | 2.73 (2.45) | 3.45 (2.21)
  BrAC = 0.04 | 3.82 (2.75) | 4.82 (3.03)
  BrAC = 0.06 | 4.45 (3.48) | 5.36 (3.33)
  BrAC = 0.08 | 5.27 (3.29) | 6.36 (2.80)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.93, ANOVA

6. Primary Outcome: Subjective Effects of Alcohol Using the Drug Effects Questionnaire (DEQ) - "Like" Subscale
Description: Subjective effects of alcohol will be measured using the Drug Effects Questionnaire, which consists of 4 items that capture subjective effects, (feeling effects, liking effects, wanting more and being high). The question "Do you like the effects you are feeling right now?" was rated on an 11 point scale from 0 to 10 (higher values represent more effects).
Time Frame: as for outcome 4
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 4.09 (1.70) | 4.09 (2.02)
  BrAC = 0.02 | 5.36 (1.63) | 5.36 (3.20)
  BrAC = 0.04 | 6.18 (2.52) | 5.55 (2.95)
  BrAC = 0.06 | 6.64 (2.98) | 6.36 (3.44)
  BrAC = 0.08 | 6.45 (3.33) | 6.27 (3.50)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.95, ANOVA

7. Primary Outcome: Subjective Effects of Alcohol Using the Drug Effects Questionnaire (DEQ) - "More" Subscale
Description: Subjective effects of alcohol will be measured using the Drug Effects Questionnaire, which consists of 4 items that capture subjective effects, (feeling effects, liking effects, wanting more and being high). The question "Would you like more of the drug right now?" was rated on an 11 point scale from 0 to 10 (higher values represent more effects).
Time Frame: as for outcome 4
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 1.64 (2.25) | 3.18 (4.00)
  BrAC = 0.02 | 4.91 (4.09) | 6.27 (4.52)
  BrAC = 0.04 | 5.45 (3.96) | 6.00 (3.95)
  BrAC = 0.06 | 5.00 (3.92) | 5.64 (4.03)
  BrAC = 0.08 | 5.27 (4.25) | 5.55 (4.78)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.43, ANOVA

8. Primary Outcome: Subjective Effects of Alcohol Using the Drug Effects Questionnaire (DEQ) - "High" Subscale
Description: Subjective effects of alcohol will be measured using the Drug Effects Questionnaire, which consists of 4 items that capture subjective effects, (feeling effects, liking effects, wanting more and being high). The question "Are you high?" was rated on an 11 point scale from 0 to 10 (higher values represent more effects).
Time Frame: as for outcome 4
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 0.91 (1.70) | 0.09 (0.30)
  BrAC = 0.02 | 2.64 (2.29) | 3.27 (2.01)
  BrAC = 0.04 | 4.00 (2.93) | 5.36 (2.66)
  BrAC = 0.06 | 4.91 (3.56) | 5.73 (2.57)
  BrAC = 0.08 | 5.09 (3.62) | 6.00 (2.79)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.06, ANOVA

9. Primary Outcome: Subjective Effects of Alcohol Using the Biphasic Alcohol Effects Scale (BAES) - Stimulant Subscale
Description: Subjective effects of alcohol will be measured using the Biphasic Alcohol Effects Scale (BAES) , which consists of 14 items designed to capture the stimulant and sedative effects of alcohol, each rated on an 11-point scale (0 = not at all, 10 = extremely). The total score for the Stimulant Subscale ranges from 0 to 70. Mean scores across all subjects are reported below.
Time Frame: as for outcome 4
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 18.09 (13.37) | 17.36 (12.99)
  BrAC = 0.02 | 20.00 (11.91) | 23.73 (14.29)
  BrAC = 0.04 | 21.73 (15.04) | 20.09 (13.32)
  BrAC = 0.06 | 25.91 (19.03) | 22.64 (15.74)
  BrAC = 0.08 | 26.18 (20.17) | 20.91 (15.00)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.21, ANOVA

10. Primary Outcome: Subjective Effects of Alcohol Using the Biphasic Alcohol Effects Scale (BAES) - Sedative Subscale
Description: Subjective effects of alcohol will be measured using the Biphasic Alcohol Effects Scale (BAES) , which consists of 14 items designed to capture the stimulant and sedative effects of alcohol, each rated on an 11-point scale (0 = not at all, 10 = extremely). The total score for the Sedative Subscale ranges from 0 to 70. Mean scores across subjects are reported below.
Time Frame: as for outcome 4
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale
  BrAC = 0.00 | 14.18 (14.67) | 10.64 (9.97)
  BrAC = 0.02 | 11.00 (13.10) | 13.09 (14.80)
  BrAC = 0.04 | 10.91 (14.72) | 16.00 (15.75)
  BrAC = 0.06 | 15.27 (17.41) | 16.73 (19.22)
  BrAC = 0.08 | 15.27 (18.93) | 16.64 (17.32)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.09, ANOVA

11. Primary Outcome: Cue-induced Craving Using the Alcohol Urge Questionnaire (AUQ)
Description: Cue-induced craving will be measured using the Alcohol Urge Questionnaire (AUQ), which consists of 8 items associated with urge to drink alcohol, rated on a 7 point scale (0 = strongly disagree, 6 = strongly agree). Item scores were averaged and the total score also ranges from 0-6.
Time Frame: 6 hours post-medication administration
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 11 | 11
scores on a scale | 3.59 (1.69) | 4.07 (1.34)
Statistical Analysis 1: Comparison: Placebo vs IVM 30mg; Test type: Superiority or Other; p = 0.99, ANOVA

12. Primary Outcome: Adverse Effects
Description: Adverse effects will be monitored to determine the safe of combining IVM (30 mg) with moderate doses of alcohol (0.08 g/dl) using the Systematic Assessment for Treatment Emergent Effects (SAFTEE). The SAFTEE is a 24-item checklist in which the participant can identify whether a symptom is present (yes/no), its severity (mild, moderate, severe) and whether it was caused by the medication (yes/no). Data below represents a count of individual adverse effects reported on the SAFTEE during the alcohol infusion.
Time Frame: During alcohol infusion at BrAC = 0.00, 0.04, 0.08 g/dl
Population: All randomized subjects included.
Measure: Number; unit: adverse effect count
Groups:
- Placebo (BrAC = 0.00): Single dose sugar pill, matched to active medication. Timepoint is at beginning of alcohol infusion when BrAC is still 0.00.
- Placebo (BrAC = 0.04): Single dose sugar pill, matched to active medication. Timepoint is during alcohol infusion when BrAC has reached 0.04.
- Placebo (BrAC = 0.08): Single dose sugar pill, matched to active medication. Timepoint is during alcohol infusion when BrAC has reached 0.08.
- IVM 30mg (BrAC = 0.00): Ivermectin (IVM): Single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin. Timepoint is at beginning of alcohol infusion when BrAC is still 0.00.
- IVM 30mg (BrAC = 0.04): Ivermectin (IVM): Single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin. Timepoint is during alcohol infusion when BrAC has reached 0.04.
- IVM 30mg (BrAC = 0.08): Ivermectin (IVM): Single dose (30 mg) of semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin. Timepoint is during alcohol infusion when BrAC has reached 0.08.
Arm/Group | Placebo (BrAC = 0.00) | Placebo (BrAC = 0.04) | Placebo (BrAC = 0.08) | IVM 30mg (BrAC = 0.00) | IVM 30mg (BrAC = 0.04) | IVM 30mg (BrAC = 0.08)
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
adverse effect count
  Abdominal pain/cramps | 0 | 1 | 1 | 0 | 0 | 0
  Yellow eyes | 0 | 0 | 0 | 0 | 0 | 0
  Nausea or vomiting | 0 | 0 | 0 | 0 | 0 | 0
  Irritability or anger | 1 | 0 | 0 | 0 | 0 | 0
  Increased desire for sex | 1 | 0 | 1 | 1 | 2 | 1
  Nervousness | 1 | 0 | 0 | 1 | 0 | 0
  Ringing in the ears | 0 | 0 | 0 | 0 | 0 | 0
  Decrease in appetite | 0 | 0 | 0 | 0 | 0 | 0
  Depression | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 1 | 2 | 2 | 1 | 1 | 2
  Difficulty in staying awake | 3 | 3 | 4 | 3 | 2 | 2
  Increase in appetite | 0 | 1 | 3 | 1 | 2 | 4
  Blurred vision | 1 | 1 | 1 | 0 | 1 | 1
  Drowsiness | 2 | 4 | 2 | 2 | 4 | 5
  Headache | 0 | 0 | 0 | 0 | 1 | 0
  Night sweats | 0 | 0 | 0 | 0 | 0 | 0
  Mental confusion | 0 | 0 | 0 | 0 | 0 | 0
  Anxiety | 0 | 0 | 0 | 0 | 1 | 0
  Joint or muscle pain | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness | 0 | 0 | 0 | 0 | 1 | 2
  Sexual problems | 0 | 0 | 0 | 0 | 0 | 0
  Difficulty sleeping | 0 | 0 | 0 | 0 | 0 | 0
  Fever or chills | 0 | 0 | 0 | 0 | 0 | 0
  Decreased desire for sex | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Ivermectin Pharmacokinetics: Peak Concentration (Cmax)
Description: This study will collect blood samples for pharmacokinetic (PK) and pharmacodynamic profiling in order to examine whether IVM metabolism corresponds to its effects on alcohol response. Maximum plasma concentration (Cmax), measured in ng/mL, provided below.
Time Frame: Hours post-drug administration: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- IVM 30mg: Ivermectin (IVM): Single dose (30 mg) of a semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum anti parasitic avermectin.
Arm/Group | IVM 30mg
Number analyzed (Participants) | 11
ng/mL | 406.03 (398.36)

14. Secondary Outcome: Ivermectin Pharmacokinetics: Time to Cmax (Tmax)
Description: This study will collect blood samples for pharmacokinetic (PK) and pharmacodynamic profiling in order to examine whether IVM metabolism corresponds to its effects on alcohol response. Time to Cmax (Tmax), measured in hours, provided below.
Time Frame: Hours post-drug administration: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IVM 30mg
Number analyzed (Participants) | 11
hours | 9.09 (3.62)

15. Secondary Outcome: Ivermectin Pharmacokinetics: Area Under the Time-concentration Curve (AUC)
Description: This study will collect blood samples for pharmacokinetic (PK) and pharmacodynamic profiling in order to examine whether IVM metabolism corresponds to its effects on alcohol response. Area under the time-concentration curve (AUC) from 0 to 48 hours after IVM administration, provided below.
Time Frame: Hours post-drug administration: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48
Population: All randomized subjects included.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | IVM 30mg
Number analyzed (Participants) | 11
ng*h/mL | 5078 (4258)

16. Secondary Outcome: Ivermectin Pharmacokinetics: Half-life (T1/2)
Description: This study will collect blood samples for pharmacokinetic (PK) and pharmacodynamic profiling in order to examine whether IVM metabolism corresponds to its effects on alcohol response. Half-life of ivermectin (T1/2), measured in hours, provided below.
Time Frame: Hours post-drug administration: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 48
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IVM 30mg
Number analyzed (Participants) | 11
hours | 15.75 (6.86)

17. Secondary Outcome: Stress-induced Alcohol Craving
Description: Alcohol Urge Questionnaire (AUQ)
Time Frame: pre-post exposure to an imaginal stress script
Population: The stress paradigm (pre-post exposure to an imaginal stress script) was not implemented from the outset of the study due to feasibility reasons. In particular, the investigators were concerned that the timing of the stress exposure might contaminate the effects of the alcohol administration.
Arm/Group | Placebo | IVM 30mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- IVM 30mg: Ivermectin 30 mg single dose
  Ivermectin: Ivermectin is a semi-synthetic macrocyclic lactone used worldwide as a broad-spectrum antiparasitic avermectin.
  Alcohol
- Placebo: Matched placebo, single dose
  Placebo: sugar pill
  Alcohol
Arm/Group | IVM 30mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No